CLINICAL TRIAL: NCT03978754
Title: Assessment of Breast Cancer-Related Arm Lymphedema-Comparison of Traditional Measurement Methods and Indocyanine Green（ICG）Lymphography
Brief Title: Assessment of Breast Cancer-Related Arm Lymphedema
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUPH18050101
Record Dates: First submitted 2019-01-23; First posted 2019-06-07 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Breast Cancer
Keywords: Lymphedema; Breast cancer; ICG lymphography; Bioelectrical impedance technology
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients who visit clinic: Postoperative patients who have undergone axillary surgery for breast cancer and went to clinic due to complaints of upper limb discomfort.（The expected number of subjects in this group is 300）
  Interventions: Diagnostic Test: ICG lymphography、CM、VD、Bioelectrical impedance technology、self-report
- Preoperative breast cancer patients: Preoperative subjects diagnosed with breast cancer were enrolled as non-lymphedema group. （The expected number of subjects in this group is 1300）
  Interventions: Diagnostic Test: Bioelectrical impedance technology、CM

INTERVENTIONS:
Diagnostic Test: ICG lymphography、CM、VD、Bioelectrical impedance technology、self-report — All of these methods are used for patients visiting the lymphedema clinic to assess whether they have developed lymphedema.
  Other Names: ICG: indocyanine green; CM: circumference measurement; VD: volume displacement
  Groups: Patients who visit clinic
Diagnostic Test: Bioelectrical impedance technology、CM — These two methods are routine evaluation methods for breast cancer patients before surgery
  Other Names: CM: circumference measurement
  Groups: Preoperative breast cancer patients

SUMMARY:
Lymphedema is a serious complication of breast cancer treatment. Reported prevalence of lymphedema following treatment for breast cancer varies, ranging from 7-45%. The reason for the wide variation in the reported incidence of lymphedema is the different measurement techniques used and the absence of an agreed diagnostic criteria. Nowadays, the common method include limb circumference measurement、volume measurement、bioimpedance spectroscopy (BIS) and self-report. Each of these methods has advantages and disadvantages. A variety of publications have demonstrated the ability of bioimpedance to diagnose subclinical lymphedema. As a new method for detecting lymphedema, some study have also shown indocyanine green（ICG）lymphography can have a certain value for the detection of subclinical lymphedema. Early detection can reduce the incidence of late-stage lymphedema in postoperative patients. Therefore, we want to explore the ability of these methods. We are going to perform baseline arm circumference measurements and bioelectrical impedance measurements for all preoperative breast cancer patients in our center. In addition, the arm circumference measurement、volume measurement、bioimpedance spectroscopy (BIS) 、self-report and indocyanine green (ICG) lymphography will be performed on patients who go to the lymphedema clinic after breast cancer surgery. First, we want to establish the threshold and reference value range based on the impedance value of patients with lymphedema and people without lymphedema.Second, we are going to examine the relationship between the most commonly used methods of lymphedema and also to test which method is more sensitive for the diagnosis of clinical and subclinical lymphedema. Finally, we want to explore the ability of ICG lymphography in detecting sub-clinical lymphedema.

DETAILED DESCRIPTION:
Breast cancer is a common malignant disease that threatens the health of women. As a serious complication of breast cancer treatment, lymphedema is caused by chronic accumulation of lymph fluid in the interstitial spaces of the affected limb or surrounding areas. Reported prevalence of lymphedema following treatment for breast cancer varies, ranging from 7-45%. One reason for the wide variation in the reported incidence of lymphedema is the different measurement techniques used and the absence of an agreed diagnostic criteria. Nowadays, the common method include limb circumference measurement、volume measurement、bioimpedance spectroscopy (BIS) and self-report. Each of these methods has advantages and disadvantages. A variety of publications have demonstrated the ability of bioimpedance to diagnose subclinical lymphedema. As a new method for detecting lymphedema, some study have also shown indocyanine green（ICG）lymphography can have a certain value for the detection of subclinical lymphedema. Early detection can reduce the incidence of late-stage lymphedema in postoperative patients. Therefore, we want to explore the ability of these methods. We are going to perform baseline arm circumference measurements and bioelectrical impedance measurements for all preoperative breast cancer patients in our center. In addition, the arm circumference measurement、volume measurement、bioimpedance spectroscopy (BIS) 、self-report and indocyanine green (ICG) lymphography will be performed on patients who go to the lymphedema clinic after breast cancer surgery.First, we want to establish the threshold and reference value range based on the impedance value of patients with lymphedema and people without lymphedema.Second, we are going to examine the relationship between the most commonly used methods of lymphedema and also to test which method is more sensitive for the diagnosis of clinical and subclinical lymphedema. Finally, we want to explore the ability of ICG lymphography in detecting sub-clinical lymphedema.

ELIGIBILITY:
The eligibility criteria for patients who visit the clinic:

Inclusion Criteria:

* Patients with breast cancer who underwent axillary surgery.
* Patients who have complaints about upper extremity lymphedema and are willing to undergo examination.
* Sign the informed consent.

Exclusion Criteria:

* Bilateral breast cancer.
* A history of allergy to contrast agents.
* There are arteriovenous thrombosis in the affected limb.
* Regional lymph node recurrence
* Did not sign informed consent.
* Serious heart, brain and other diseases.
* The primary lymphatic system diseases (such as lymphatic leakage).
* Only one side of the limb received ICG angiography.

The eligibility criteria for preoperative subjects diagnosed with breast cancer:

Inclusion Criteria:

• Preoperative subjects diagnosed with breast cancer at our breast center.

Exclusion Criteria:

• We strictly excluded all possible causes of lymphedema. Subjects whose clinical stage of lymph node is N2 or higher were excluded. Subjects with lymphedema -related diseases or kidney disease, inflammatory breast cancer, a history of axillary surgery, radiotherapy to the upper limbs or the chest wall, soft tissue infection, pregnancy, congestive heart-failure, administration of diuretics (which may have significantly changed the hydration status) and implanted devices (e.g., pacemakers), were also excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group1: Patients who visit the clinic; Group2: Preoperative subjects diagnosed with breast cancer.
Sampling Method: Non-Probability Sample
Enrollment: 1600 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of indocyanine green (ICG) lymphography | 2017-2022
  Sensitivity means the ability of detecting patients with true lymphedema. Specificity means the ability of detecting non-lymphedema patients.
The incidence of lymphedema | 2017-2022
  The incidence of lymphedema assessed by different methods when patients first visit clinic
The cutoff value of BIS | 2017-2022
  studies on the threshold value established by Inbody 720 device have been extremely limited. We aimed to determine its reference range and cutoff values.
The occurrence of lymphedema after follow-up | 2017-2022
  Patients who don't develop lymphedema when the first visit to the lymphedema clinic, the occurrence of lymphedema after follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Wang Shu, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Azhar SH, Lim HY, Tan BK, Angeli V. The Unresolved Pathophysiology of Lymphedema. Front Physiol. 2020 Mar 17;11:137. doi: 10.3389/fphys.2020.00137. eCollection 2020. PMID 32256375
- [Background] Executive Committee of the International Society of Lymphology. The diagnosis and treatment of peripheral lymphedema: 2020 Consensus Document of the International Society of Lymphology. Lymphology. 2020;53(1):3-19. PMID 32521126
- [Background] Czerniec SA, Ward LC, Refshauge KM, Beith J, Lee MJ, York S, Kilbreath SL. Assessment of breast cancer-related arm lymphedema--comparison of physical measurement methods and self-report. Cancer Invest. 2010 Jan;28(1):54-62. doi: 10.3109/07357900902918494. PMID 19916749
- [Background] Qin ES, Bowen MJ, Chen WF. Diagnostic accuracy of bioimpedance spectroscopy in patients with lymphedema: A retrospective cohort analysis. J Plast Reconstr Aesthet Surg. 2018 Jul;71(7):1041-1050. doi: 10.1016/j.bjps.2018.02.012. Epub 2018 Apr 9. PMID 29650264
- [Background] Yamamoto T, Yamamoto N, Doi K, Oshima A, Yoshimatsu H, Todokoro T, Ogata F, Mihara M, Narushima M, Iida T, Koshima I. Indocyanine green-enhanced lymphography for upper extremity lymphedema: a novel severity staging system using dermal backflow patterns. Plast Reconstr Surg. 2011 Oct;128(4):941-947. doi: 10.1097/PRS.0b013e3182268cd9. PMID 21681123
- [Background] Akita S, Nakamura R, Yamamoto N, Tokumoto H, Ishigaki T, Yamaji Y, Sasahara Y, Kubota Y, Mitsukawa N, Satoh K. Early Detection of Lymphatic Disorder and Treatment for Lymphedema following Breast Cancer. Plast Reconstr Surg. 2016 Aug;138(2):192e-202e. doi: 10.1097/PRS.0000000000002337. PMID 27465179
- [Background] Ward LC. Bioelectrical impedance analysis: proven utility in lymphedema risk assessment and therapeutic monitoring. Lymphat Res Biol. 2006 Spring;4(1):51-6. doi: 10.1089/lrb.2006.4.51. No abstract available. PMID 16569209
- [Background] Fu MR, Cleland CM, Guth AA, Kayal M, Haber J, Cartwright F, Kleinman R, Kang Y, Scagliola J, Axelrod D. L-dex ratio in detecting breast cancer-related lymphedema: reliability, sensitivity, and specificity. Lymphology. 2013 Jun;46(2):85-96. PMID 24354107
- [Background] Ward LC, Czerniec S, Kilbreath SL. Quantitative bioimpedance spectroscopy for the assessment of lymphoedema. Breast Cancer Res Treat. 2009 Oct;117(3):541-7. doi: 10.1007/s10549-008-0258-0. Epub 2008 Dec 11. PMID 19082708